CLINICAL TRIAL: NCT06416254
Title: The Effects of a Diet Enriched With Dietary Fibre on Glycaemic Response, Gastrointestinal Tolerability, Satiety, and Microbiome Functionality (The Fibre Full Study).
Brief Title: The Fibre Full Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: APC170
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Overweight and Obesity
Keywords: Dietary fiber; glycemic control; gastrointestinal microbiome; microbiota; overweight; obesity; metabolism; satiety
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Crossover: Participants receive one of two (or more) alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibre-enriched (Active Comparator): During the fibre-enriched arm, participants will receive the fibre-rich diet containing fibre-enriched foods provided through a full meal plan to be consumed throughout the day.
  Interventions: Other: Fibre-enriched diet
- Control (Placebo Comparator): During the control arm, participants will receive a non-fibre enriched diet consisting of matched control foods provided through a full meal plan otherwise identical to the fibre-enriched arm.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Fibre-enriched diet — The fibre-enriched diet contains fibre-enriched foods in which a portion of digestible carbohydrates are replaced with isolated dietary fibres. The fibre-enriched study foods are consumed as part of a full meal plan provided to participants.
  Arms: Fibre-enriched
Other: Control diet — The control diet contains non-fibre-enriched study foods. The control study foods are consumed as part of a full meal plan provided to participants.
  Arms: Control

SUMMARY:
This study will systematically investigate the effects of a diet with decreased energy density, reduced glycaemic index, and significantly increased dietary fibre, on post-prandial glycaemic response, satiety, gastrointestinal tolerability and gut microbiota composition and function in individuals with excess body weight (Body Mass Index (BMI) 25-35kg/m2).

Hypothesis: The investigators hypothesise that a diet enriched in fibre will be beneficial to post-prandial glycaemic response, well tolerated and satiating, as compared to the standard Western-style diet.

DETAILED DESCRIPTION:
Participants: Healthy men and pre-menopausal, non-pregnant and non-lactating women, 18-45 years of age, with a Body Mass Index (BMI) between 25-34.9 kg/m2 will be recruited (n=20).

Study Design: This exploratory study aims to investigate the effects of a fibre-enriched (FR) diet in adults with excess body weight in comparison to a control diet. This randomized, single-blinded, placebo-controlled intervention/trial with a crossover design compares the effects of consumption of fibre-enriched food staples delivered within a full meal plan (fibre-enriched diet plan) with a matched control meal plan (control diet plan).

Participants stratified by age and BMI, will be randomly assigned to receive either the control diet or fibre-enriched (FR) diet for 8 days. After these 8 days, a washout period (13 day minimum) will commence, and participants will then crossover to the opposite diet. All foods and prepared meals within the menu plan will be provided to participants for both the control and FR diets. Participants are required to strictly adhere to their assigned meal plan for the 8-day period.

Given the higher dietary fibre intake of the FR-diet, the study design incorporates a dose escalation of the fibre content to allow participants on the FR diet to adjust to the increase in dietary fibre intake (4-day reduced dose, wherein study foods contain only a portion of the required dose of fibre, and 4-day full dose, high fibre intake).

The effect of the FR diet on satiety and overall food intake will be assessed. Participants on the FR diet and the control diet will be provided with non-fibre enriched snacks which they may consume at designated times each day, if they wish to and in ab libitum. These snacks will be an optional component of the menu plan. All food intakes will be monitored, and all leftovers will be returned to the research team. Additionally, dietary assessments will be completed at regular intervals.

Study Treatments:

* The FR diet consists of a full meal plan containing engineered common food products with decreased energy density and glycaemic index, in which a large proportion of refined carbohydrates are replaced with dietary fibre.
* The control diet consists of a full meal plan with non-fibre enriched food products.

Study Outcome measures will include post-prandial glycaemic response, satiety, gastrointestinal tolerability and gut microbiota composition and function in individuals with excess body weight (BMI 25-35kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to give written informed consent.
* Be between 18 and 45 years of age
* Have a Body Mass Index (BMI) of 25-34.9kg/m2 (Overweight or Obese Class I)
* Have had a stable body weight (≤5% change over the past three months)
* Be in general good health as determined by the investigator through interview and vital signs (blood pressure, pulse, temperature). Systolic blood pressure less than 160mm Hg and diastolic blood pressure less than 100 mm Hg (defined as Hypertension stage 2).
* Be willing to avoid consuming dietary supplements, prebiotics, probiotics, or fibre-rich supplements within four weeks prior to the baseline visit, and until the end of the study.
* Be willing to avoid physical exercise for the duration of the study (physical exercise defined as any physical activity that is planned to achieve a fitness goal)
* Be willing to consume the investigational products daily for the duration of the study.

Exclusion Criteria:

* Pregnant, lactating, menopausal or post-menopausal women, or women who are planning to become pregnant over the study period.
* Have had antibiotic treatment within three months prior to baseline.
* Are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of study results; to include: anti-inflammatory drugs, H2 blockers, antacid, proton pump inhibitors, anti-hypertensive medications, corticosteroids, laxatives, enemas, antibiotics, anti-coagulants, immunosuppressant medication. Participants should have a wash-out period of at least two-weeks for each of these medications except for antibiotics, which should not have been taken in the previous three months. Participants taking proton pump inhibitors and medications for chronic conditions (e.g., anti-hypertensive medication) will be allowed onto the study if the dose has been stable for at least two months prior to the study baseline visit.
* Have a history or indication of drug and/or alcohol abuse at the time of enrolment.
* Have a habitual alcohol consumption of >2 alcoholic beverages/day (>28g ethanol daily).
* Follow a vegetarian or vegan diet
* Have a typical fibre intake of >30g per day
* Have experienced major dietary changes within three months prior to the study baseline.
* Plan major lifestyle changes (diet, physical activity, or travel) during the study period.
* Have a clinically diagnosed eating disorder.
* Have a food allergy or intolerance that would preclude study product intake (for example eggs, gluten, nuts, milk or any other food allergy or intolerance)
* Have an active gastrointestinal disorder or previous gastrointestinal surgery
* Have a significant active and medically-diagnosed acute or chronic co-existing illness including: metabolic, psychiatric, cardiovascular, endocrinological, immunological condition, gastrointestinal disease or any other condition which contraindicates, in the investigator's judgement, entry to the study (such as, diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis A/B/C, HIV, cancer, diabetes etc) or a significant history of such diseases.
* Are severely immunocompromised (e.g., HIV positive, transplant patient, on anti-rejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last 12 months).
* Have a malignant disease or concomitant end-stage organ disease.
* Have symptomatic respiratory or cardiac illness.
* Experience alarm features such as sudden weight loss, rectal bleeding, a recent change in bowel habits, or significant abdominal pain within three months prior to baseline.
* Individuals who, in the opinion of the investigator are poor attendees or unlikely for any reason to be able to comply with the study protocol.
* Participants may not be receiving treatment involving experimental drugs.
* If the participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Individuals with pacemakers or implantable cardioverter defibrillators.
* Individuals that regularly undertake rigorous exercise, defined by International Physical Activity Questionnaire with a score within category 3, Health Enhancing Physical Activity (HEPA) Active.
* Individuals who smoke or vape regularly (i.e., daily or habitual use).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — An equal number of male and female participants will be enrolled
Enrollment: 20 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Impact of a fibre-enriched diet on glycaemic control | Assessments will be conducted continuously over each 8-day intervention period
  Changes in glycaemic response using continuous interstitial glucose monitoring when consuming the fibre-enriched diet compared to a matched control diet.
Differences in participant reported satiety when consuming the fibre-enriched diet compared to the matched control diet | Throughout each 8-day intervention period assessed at specific time points during the day (e.g. pre- and post-meal consumption)
  Differences in satiety assessed by analysis of Participant responses to the Satiety Labelled Intensity Magnitude (SLIM) scale and assessment of food consumption. The SLIM scale assesses perceived hunger/fullness using 11 phrases placed along a vertical line scale with "Greatest imaginable hunger" (score = -100) at the bottom and "Greatest imaginable fullness" at the top (score = +100).

SECONDARY OUTCOMES:
Gastrointestinal tolerance to dietary fibre assessed by a Gastrointestinal Symptom and Bowel Movement Questionnaire | Throughout each 8-day intervention period, assessed at specific time points (i.e. at baseline, 4 days (mid-point) and 8 days (end) of each dietary intervention)
  Evaluation of the impact of the fibre-enriched diet on gastrointestinal tolerance, through monitoring of participant reported gastrointestinal symptoms. This will be assessed via a Gastrointestinal Symptom and Bowel Movement Questionnaire comprising eleven questions from The Gastrointestinal Symptom Rating Scale (GSRS) followed by the Bristol Stool Chart and bowel frequency and flatus questions. The GSRS utilizes a 7-point response scale to measure the level of discomfort associated with a given gastrointestinal symptom, ranging from "No discomfort at all" to "Very severe discomfort." Participants will also rate the form of their stool sample using the Bristol Stool Chart.
Impact of a fibre-enriched diet on gut microbiota composition | Assessments may be conducted at baseline (pre-intervention), and then at 4 days (mid-point) and 8 days (end) of each study intervention period.
  Changes in gut microbiome composition and diversity between intervention periods through 16S ribosomal RNA (rRNA) gene sequencing of faecal samples.
Effect of a fibre-enriched diet on gut microbiota function | Assessments may be conducted at baseline (pre-intervention), and then at 4 days (mid-point) and 8 days (end) of each study intervention period.
  Changes in faecal metabolite concentrations determined through liquid chromatography-mass spectrometry (LC-MS)

OTHER OUTCOMES:
Impact of a fibre-enriched diet on gut inflammatory marker concentration. | Assessments may be conducted at baseline (pre-intervention), and then at the end of each 8 day intervention period.
  Changes in gut inflammatory marker concentration using established methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Walter, PhD, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armet AM, Deehan EC, Thone JV, Hewko SJ, Walter J. The Effect of Isolated and Synthetic Dietary Fibers on Markers of Metabolic Diseases in Human Intervention Studies: A Systematic Review. Adv Nutr. 2020 Mar 1;11(2):420-438. doi: 10.1093/advances/nmz074. PMID 31342059
- [Background] Baenziger PS, Frels K, Greenspan S, Jones J, Lovegrove A, Rose D, Shewry P, Wallace R. A stealth health approach to dietary fibre. Nat Food. 2023 Jan;4(1):5-6. doi: 10.1038/s43016-022-00674-w. No abstract available. PMID 37118563
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Deehan EC, Walter J. The Fiber Gap and the Disappearing Gut Microbiome: Implications for Human Nutrition. Trends Endocrinol Metab. 2016 May;27(5):239-242. doi: 10.1016/j.tem.2016.03.001. Epub 2016 Apr 11. PMID 27079516
- [Background] Hall KD, Ayuketah A, Brychta R, Cai H, Cassimatis T, Chen KY, Chung ST, Costa E, Courville A, Darcey V, Fletcher LA, Forde CG, Gharib AM, Guo J, Howard R, Joseph PV, McGehee S, Ouwerkerk R, Raisinger K, Rozga I, Stagliano M, Walter M, Walter PJ, Yang S, Zhou M. Ultra-Processed Diets Cause Excess Calorie Intake and Weight Gain: An Inpatient Randomized Controlled Trial of Ad Libitum Food Intake. Cell Metab. 2019 Jul 2;30(1):67-77.e3. doi: 10.1016/j.cmet.2019.05.008. Epub 2019 May 16. PMID 31105044
- [Background] Ludwig DS, Ebbeling CB. The Carbohydrate-Insulin Model of Obesity: Beyond "Calories In, Calories Out". JAMA Intern Med. 2018 Aug 1;178(8):1098-1103. doi: 10.1001/jamainternmed.2018.2933. PMID 29971406
- [Background] Rouhani MH, Haghighatdoost F, Surkan PJ, Azadbakht L. Associations between dietary energy density and obesity: A systematic review and meta-analysis of observational studies. Nutrition. 2016 Oct;32(10):1037-47. doi: 10.1016/j.nut.2016.03.017. Epub 2016 Mar 31. PMID 27238958
- [Background] Sonnenburg ED, Sonnenburg JL. Starving our microbial self: the deleterious consequences of a diet deficient in microbiota-accessible carbohydrates. Cell Metab. 2014 Nov 4;20(5):779-786. doi: 10.1016/j.cmet.2014.07.003. Epub 2014 Aug 21. PMID 25156449
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418